CLINICAL TRIAL: NCT06468072
Title: Exploring the Impact of Theatrical Expressive Tasks in Children With Autism Spectrum Disorder (ASD).
Brief Title: Exploring Theatrical Expressive Tasks for Children With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-008
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: autism; children; expressiveness; theater; technology
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with autism (Experimental): The experimental group consists of 10 children diagnosed with autism who voluntarily attend the CNR-IRIB in Messina. The sample is aged between 7 and 11 years with severity level 1 (minimum support required)
  Interventions: Other: Expressivity protocol for children with autism
- Non-autistic children (Other): The comparison group consists of 10 non-autistic children with no other diagnosis, who voluntarily attend the CNR-IRIB in Messina. The sample is between 7 and 11 years old.
  Interventions: Other: Expressivity protocol for non-autistic children

INTERVENTIONS:
Other: Expressivity protocol for children with autism — The activities proposed by this protocol stimulate different expressive skills, which are often lacking in people with autism. For this reason, the protocol is based on the strengthening of the following skills: perception of the body in movement in the space (4 sessions), the expressiveness of the body in its entirety (4 sessions), breathing and the use of the voice to express emotions in relation to the environment (4 sessions), rhythm and movement, to develop motor coordination and the expressiveness of movements (4 sessions). The protocol consists of 16 sessions: a weekly group session lasting one hour.
  Arms: Children with autism
Other: Expressivity protocol for non-autistic children — The activities proposed by this protocol stimulate different expressive skills. The protocol is based on the strengthening of the following skills: perception of the body in movement in space (4 sessions), the expressiveness of the body in its entirety (4 sessions), breathing and the use of the voice to express emotions in relation to the environment (4 sessions), rhythm and movement, to develop motor coordination and the expressiveness of movements (4 sessions). The protocol consists of 16 sessions: a weekly group session lasting one hour.
  Arms: Non-autistic children

SUMMARY:
Autism Spectrum Disorder (ASD), according to the diagnostic criteria of Diagnostic and Statistical Manual of Mental Disorders- V Edition (DSM-5), is a disorder involving (a) persistent deficits in social communication, social interaction and (b) patterns of restricted and stereotyped behavior and/or interests and/or activities. Specifically, impairment in social interaction manifests itself in different areas of individual functioning and through various facets: social-emotional reciprocity, poor understanding of social rules, reduced sharing of interests, emotions or feelings, reduced or absent theory of mind, inability to initiate or respond to social interactions (turn-taking in conversation), and difficulties in the use of communication. Facial expressions, vocal intonation, postures and gestures are crucial components of non-verbal communication that play a fundamental role in social-communicative functions. However, people with ASD may show significant deficits in these forms of expression, negatively affecting the ability to generate an appropriate social response, which is essential for initiating and maintaining social interactions. Children with ASD tend to avoid eye contact with others and show little or no interest in people, often looking past them or away from them. This behavior contributes to presenting them as "markedly aloof and distant". The aim of the study is to explore the effect of specific expressive tasks, conducted by highly qualified personnel, in a group setting, by means of targeted theatrical activities. These activities include exercises focusing on the use of voice and posture, the variety of vocal intonations and the harmonization between verbal production and facial expressiveness. In the context of this study, 20 children will be involved, divided into an experimental group and a control group. The experimental group will include 10 children with ASD who voluntarily participate in activities organized by the IRIB-CNR of Messina. These children, aged between 6 and 11 years, present a medium-high level of cognitive functioning, as assessed by the Wechsler Intelligence Scale for Children- IV Edition (WISC-IV) cognitive test. In parallel, the control group will consist of 10 normo-typical children, selected from the Istituto Comprensivo San Francesco di Paola of Messina, having the same age group, who will not participate in the experimental activities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder;
* Age between 6 and 11 years;
* IQ over 80 assessed by means of WISC-IV.

Exclusion Criteria:

* Presence of other medical disorders

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Profiling Elements of Prosodic Systems in Children (PEPS-C) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change.
  Profiling Elements of Prosody in Speech-Communication (PEPS-C) is a semi-automated test battery for assessing receptive and expressive prosody skills. It has been used in several studies of the speech and understanding of children with high-functioning autism/Asperger's syndrome (see Prosody and autism spectrum conditions). It is intended for use by language teachers, clinicians and researchers in assessing prosody in any conditions in both children and adults.
  PEPS-C comprises 14 tasks, addressing receptive and expressive skills in parallel. The tasks are at two levels, examining prosodic function and prosodic form respectively. The assessment of skills at two levels helps to determine the level at which a testee has a problem with prosody, thus enabling better targeting of intervention. The range score is min 0 -max 192.
Pragmatic Skills in the Medea Language (APL MEDEA) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change
  APL Medea is an assessment battery for pragmatic language skills developed at the Cognitive Psychology and Neuropsychology Service of the IRCCS 'Eugenio Medea'.
  Structure:
  Metaphors (M), divided into Verbal Metaphors (MV) and Figurative Metaphors (MF): investigates the ability to understand metaphorical language.
  Comprehension of implicit meaning (CSI): assesses the ability to draw inferences about non-explicit content, range scores min 0 -max 72.
  Comics (F): assesses the ability to understand and respect the dialogic structure in a communication, range scores min 0 -max 72.
  Situations (S): assesses the ability to understand and appropriate the meaning assumed by particular expressions in social interaction, range scores min 0 -max 72.
  The Colour Game (GC): assesses the ability to use language in a referential manner and use skills related to "Theory of Mind", range scores min 0 -max 72.
Test for understanding emotions (TEC) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change.
  This test assesses the presence and development of emotional competence in children aged 3 to 11 years.
  The test consists of 23 numbered cardboard plates. The first five boards depict four different emotional expressions each, alternating randomly. For each of them, the child is asked to identify a specific emotion. The structure of the remaining boards is instead unique: for each component, the upper part of the board represents a small story with emotional content, where the face of the protagonist is left blank. The lower part, represents four different emotional expressions, from which the child is asked to choose the corresponding one. The administration is individual.
  From the application of the instrument, the authors came to the identification of a meta-emotional competence divided into three developmental areas categorisation of emotions in relation to their nature, understanding of the causes of emotions, control of emotions. The range score is min -0,3 - max 3,78.
Movement Assessment Battery for Children - Second Edition (ABC-Movement - 2) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change.
  The Movement ABC-2 battery identifies and describes the movement difficulties of children and adolescents from 3 to 16 years of age. The battery enables assessment and intervention planning in line with the bio-psycho-social model of human functioning. The Movement ABC-2 battery consists of 3 components:
  A standardized test consisting of 24 tests divided into groups of 8 tasks for 3 age groups (3-6; 7-10; 11-16), for 3 competence areas (Manual Dexterity, Aiming and Grasping, Balance). In addition to the total score, it is also possible to obtain separate scores for the three competence areas. The range score is min 1- max 19.
  An observational checklist consisting of 43 items divided into three sections, it must be completed by an adult who has the opportunity to observe the child in his/her daily motor activities.
  A manual checklist that describes the ecological approach to intervention for children with movement difficulties.
Children's Communication Checklist - Second Edition (CCC-2) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change.T
  The CCC-2 is a test that assesses the presence of communicative problems of a pragmatic nature that are difficult to assess with traditional tests. It consists of 70 multiple-choice items divided into 10 scales each containing seven items. For each scale, five items describe difficulties and two items describe strengths. The respondent is asked to rate the frequency with which different behaviors occur.
  The scales are as follows: Eloquence, Syntax, Semantics, Coherence, Inappropriate beginning, Stereotyped language, Use of context, Non-verbal communication, Social relations, Interests (range score min 1 - max 280) Using these scales, two global scores can be calculated, the Global Communication Score (GCC) and the Global Social Interaction Discrepancy Score (SIDC).
  The questionnaire is completed by an adult who has regular contact with the child or young person, preferably a parent.
Social Responsiveness Scale (SRS) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change.
  The SRS assesses reciprocal social behavior, communication and repetitive and stereotyped behavior characteristic of autism spectrum disorders in subjects between 4 and 18 years.
  A total score gives a measure of the severity of the social deficit and allows comparisons between different settings and assessors. The SRS is divided in the following subscales.
  Social awareness: ability to pick up social cues (range scores min 30- max ≥ 90).
  Social cognition: ability to interpret social signals once they have been perceived (range scores min 30-max ≥ 90).
  Social communication: includes expressive social communication (range scores min 30-max ≥ 90).
  Social motivation: indicates the extent to which a subject is generally motivated to engage in social-interpersonal behavior (range scores min 30-max ≥ 90).
  Autistic mannerisms: include stereotyped behavior or highly restricted interests characteristic of autism (range scores min 30-max ≥ 90).
Khymeia Virtual Reality Rehabilitation System (VRRS) | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change.
  Advanced software for analyzing facial expressions, it allows artificial intelligence technologies to accurately identify and interpret a broad spectrum of human emotions, recording facial movements, including those of the mouth, eyes and eyebrows, as well as the static balance of each child participating in the study.
NEuroPSYcology second edition (NEPSY-II) evaluations | The test will be scheduled pre intervention (T0) and at the study conclusion, about 1 year (T1). The T0 and T1 evaluations were conducted to determine whether the protocols carried out made a change. The test needs about 120-180 minutes.
  Secondary Outcome Measure Description. NEuroPSYcology second edition (NEPSY-II) is the most internationally known battery for assessing neuropsychological development in developmental age. Each NEPSY-II test provides raw scores that must be converted into scalar scores (min 1 - max 19) or percentile scores (min <2% - max >75%) according to the conversion tables in the manual. Neuropsychology II Edition (NESPY)' s Theory of Mind (ToM) subtest, section A is used in this protocol. Assesses the ability to decode and interpret others' intentions and life points and understand how they influence behavior. The test will be given to children pre- and post-intervention.
  The ToM test is divided into verbal: the child is read scenarios or shown figures and asked questions that require understanding of the other's point of view; nonverbal: the child is asked to choose the emotional expression appropriate to the mood of a character depicted in certain contexts.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanchi, P., Peppé, S., & Zampini, L. (2022). Prosodic development from 4 to 10 years: Data from the Italian adaptation of the PEPS-C. Speech Communication, 144, 10-19. https://doi.org/10.1016/j.specom.2022.08.007
- [Background] Lord C, Elsabbagh M, Baird G, Veenstra-Vanderweele J. Autism spectrum disorder. Lancet. 2018 Aug 11;392(10146):508-520. doi: 10.1016/S0140-6736(18)31129-2. Epub 2018 Aug 2. PMID 30078460
- [Background] Mandy W, Wang A, Lee I, Skuse D. Evaluating social (pragmatic) communication disorder. J Child Psychol Psychiatry. 2017 Oct;58(10):1166-1175. doi: 10.1111/jcpp.12785. Epub 2017 Jul 25. PMID 28741680
- [Background] Paul, R., & Simmons, E. (2019). Communication and its development in autism spectrum disorders. In Autism and Pervasive Developmental Disorders.